CLINICAL TRIAL: NCT06580626
Title: Decompression Technique Versus Ridge Splitting and Ethoss Bone Regeneration in Horizontal Ridge Augmentation With Simultaneous Implant Placement
Brief Title: Various Techniques of Horizontal Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elsheikh, assistant professor of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0108024OS
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- decompression group (Experimental)
  Interventions: Procedure: decompression technique
- Ethoss group (Experimental)
  Interventions: Procedure: guided bone regenaration using Ethoss
- ridge splitting group (Experimental)
  Interventions: Procedure: ridge splitting technqiue

INTERVENTIONS:
Procedure: decompression technique — 14 implants will be placed in patients of missing single tooth or multiple teeth in posterior mandible with subsequent horizontal ridge augmentation by decompression technique.
  Arms: decompression group
Procedure: guided bone regenaration using Ethoss — 14 implants will be placed in patients of missing single tooth or multiple teeth in posterior mandible with subsequent horizontal ridge augmentation by guided bone regeneration using β-TCP/CS synthetic bone substitute.
  Arms: Ethoss group
Procedure: ridge splitting technqiue — 14 implants will be placed in patients of missing single tooth or multiple teeth in posterior mandible with subsequent horizontal ridge augmentation by ridge splitting technique using piezosurgery.
  Arms: ridge splitting group

SUMMARY:
42 patients will be selected from the Outpatient Clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University for replacement of missed single tooth or multiple teeth in posterior mandible by dental implant in horizontally atrophic ridge.

ELIGIBILITY:
Inclusion Criteria:

* Patient's cooperation, motivation and good oral hygiene.
* Patient medically free from systemic diseases that absolutely contraindicate implant surgery.
* Moderately atrophic posterior mandibular alveolar ridge width (more than 4 mm), with minimum 10 mm height.
* Free from history of bruxism / parafunctional habits.

Exclusion Criteria:

* Patients with local pathological disease such as cyst, tumor at the planned surgical site.
* Pregnant patients.
* Heavy smoker patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width. | 1 year
  Overall width of the ridge was evaluated preoperatively, after implant placement immediately, after 6, and 12 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No